CLINICAL TRIAL: NCT02422589
Title: A Phase I, Multi-center, Open Label, Drug-drug Interaction Study to Assess the Effect of Ceritinib on the Pharmacokinetics of Warfarin and Midazolam Administered as a Two-drug Cocktail in Patients With ALK-positive Advanced Tumors Including Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase I, Multi-center, Open Label, Drug-drug Interaction Study to Assess the Effect of Ceritinib on the Pharmacokinetics of Warfarin and Midazolam in Patients With ALK-positive Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLDK378A2103; 2014-003741-95 (EudraCT Number)
Record Dates: First submitted 2015-03-16; First posted 2015-04-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2019-07

CONDITIONS: ALK-positive Advanced Tumors
Keywords: ALK-positive advanced tumors; midazolam; warfarin; ceritinib; ALK; CYP3A-4; Drug drug intereaction
MeSH Terms: interventions — ceritinib; Warfarin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ceritinib (Experimental)
  Interventions: Drug: ceritinib; Drug: warfarin; Drug: midazolam

INTERVENTIONS:
Drug: ceritinib
Drug: warfarin
Drug: midazolam

SUMMARY:
The purpose of this study was to evaluate the potential inhibitory effects of ceritinib on the CYP3A4- and CYP2C9-mediated metabolism of the probe drugs midazolam and warfarin, respectively, when administered simultaneously as a cocktail. The results obtained from this drug interaction study would provide guidance that would enable an update to the ceritinib labeling and ouldl help guide recommendations for administration of co-medications in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed diagnosis of stage IIIB (and is not a candidate for definitive multimodality therapy) or stage IV NSCLC demonstrated ALK-positive or an advanced tumor, other than NSCLC, that carries an ALK genetic alteration (mutation, translocation or amplification) and/or ALK overexpression that has progressed despite standard therapy, or for which no effective standard therapy exists.

* The test to confirm ALK-positivity may be performed in archival tumor (obtained at or since the time of diagnosis), or in a newly obtained tumor sample taken prior to the first day of study drug. Results confirming ALK-positive status must be available before initiating treatment with ceritinib.
* Patients who have received prior chemotherapy, other ALK inhibitors, biologic therapy, or other investigational agents, must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (CTCAE v 4.03) prior to starting study drug. Patients with grade ≤ 2 peripheral neuropathy or any grade of alopecia, nail changes or skin changes are allowed to enter the study.
* Patients who have been treated with chemotherapy, with biological therapy or other investigational agent must have discontinued the treatment at least 2 weeks (14 days) prior to starting the study drug on Study Day 1.In case last chemotherapy contained nitrosourea or mitomycin C, the treatment was discontinued at least 6 weeks prior to starting study drug.
* Patient has the ability to understand and provide signed informed consent.

Exclusion Criteria:

* Patients with known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate), midazolam and warfarin as described in the local product information.
* History of carcinomatous meningitis.
* Presence or history of a malignant disease other than an ALK-positive advanced tumor that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
* Clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:
* Unstable angina within 6 months prior to screening.
* Myocardial infarction within 6 months prior to screening.
* History of documented congestive heart failure (New York Heart Association functional classification III-IV).
* Uncontrolled hypertension defined by a Systolic Blood Pressure ≥ 160 mmHg and/or Diastolic Blood Pressure ≥ 100 mmHg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication (s) was allowed prior to screening.
* Ventricular arrhythmias.
* Supraventricular and nodal arrhythmias not controlled with medication.
* Other cardiac arrhythmia not controlled with medication.
* Corrected QT (QTcF) > 470 ms using Fridericia's correction on the screening electrocardiogram (ECG) (as mean of triplicate ECGs).
* Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100 mmHg, with or without anti-hypertensive medication.
* Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).

Other Protocol defined Inclusion/Exclusion may applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Phamacokinetics (PK) parameters of probe drugs and their metabolites in the absence or presence of ceritinib dosing, including but not limited to: AUCinf | Days 1,2,3,4,5,6,7,28,29,30,31,32,33,34 and once every 21 days until death or up to 24 months.
PK parameters of probe drugs and their metabolites in the absence or presence of ceritinib dosing, including but not lastlimited to: AUC | Days 1,2,3,4,5,6,7,28,29,30,31,32,33,34 and once every 121 days until death or up to 24 months.
PK parameters of probe drugs and their metabolites in the absence or presence of ceritinib dosing, including but not lastlimited to:Cmax | Days 1,2,3,4,5,6,7,28,29,30,31,32,33,34 and once every 21 days until death or up to 24 months.
PK parameters of probe drugs and their metabolites in the absence or presence of ceritinib dosing, including but not lastlimited to:Tmax | Days 1,2,3,4,5,6,7,28,29,30,31,32,33,34 and once every 21 days until death or up to 24 months.

SECONDARY OUTCOMES:
Ctrough concentrations of ceritinib | Days 1,2,3,4,5,6,7,28,29,30,31,32,33,34 and once every 21 days until death or up to 24 months.
Number of participants with Adverse Events as a measure of safety and tolerability | Days 1,2,3,4,5,6,7,28,29,30,31,32,33,34 and once every 21 days until death or up to 24 months.
  This will be done by looking at the vital signs, lab values and ECG
Objective Response Rate (ORR) | Baseline, every 6 weeks until week 27
  Tumor evaluation will be determined locally by investigator per RECIST 1.1
Duration of Response (DOR) | Baseline, every 6 weeks until week27
  Tumor evaluation will be determined locally by investigatorper RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (3):
  - Karmanos Cancer Institute Oncology Department, Detroit, Michigan
  - Henry Ford Hospital SC, Detroit, Michigan
  - Cancer Therapy & Research Center UT Health Science Center SC-4, San Antonio, Texas
- Novartis Investigative Site, Copenhagen, Denmark
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Padua, PD
- Spain (2):
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLDK378A2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17277